CLINICAL TRIAL: NCT01239745
Title: A Non-Interventional Study With Aromasin® As Adjuvant Treatment In Postmenopausal Women With Invasive, Estrogen Receptor Positive Early Breast Cancer Who Are Disease-Free After 2-3 Years Of Initial Adjuvant Tamoxifen Therapy
Brief Title: Aromasin® As Adjuvant Treatment In Postmenopausal Women With Invasive, Estrogen Receptor Positive Early Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5991094
Record Dates: First submitted 2010-11-03; First posted 2010-11-11 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Breast Neoplasms
Keywords: Hormone adjuvant treatment of early breast cancer with aromatase inhibitors following 2-3 years of tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Aromasin

INTERVENTIONS:
Drug: Aromasin — Aromasin® one 25 mg tablet to be taken once daily
  Other Names: Exemestane

SUMMARY:
This non-interventional study will be conducted in several Eastern European countries to assess the safety, tolerability and efficacy of Aromasin® when it is administered in real-word setting in postmenopausal women with invasive estrogen receptor positive early breast cancer , who are disease-free after completion of 2 to 3 years of tamoxifen and continue the treatment with Aromasin® until completion of 5 years of adjuvant hormonal therapy, to understand how Aromasin® is used in routine clinical practice, to assess adherence to prescribed Aromasin® treatment and to understand reasons for its early discontinuation.

DETAILED DESCRIPTION:
The study prematurely discontinued on October 11, 2011 due to slow enrollment. It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females, defined as one from the next :

  1. Natural menopause ≥1 year,
  2. Surgical ovariectomy,
  3. Chemotherapy-induced amenorrhoea ≥ 2 years.
* Patients who have had surgical treatment for histologically confirmed breast cancer that was non-metastatic at the time of the initial diagnosis.
* Patients who are disease-free after 2 to 3 years of adjuvant tamoxifen treatment.
* Patients whose tumour was estrogen receptor positive (ER+).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients for whom Aromasin® treatment is contraindicated (see SmPC).
* Metastatic breast cancer or a contra lateral tumour.
* Other concomitant adjuvant endocrine therapy.
* Other concomitant antineoplastic treatment.
* Participation in a clinical trial with an investigational drug during the 30 days prior to enrolment in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Estrogen receptor positive early breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Croatia (8):
  - General Hospital Karlovac, Karlovac
  - University Hospital Center Osijek, Osijek
  - General Hospital Pula, Pula
  - University Hospital Center Rijeka, Rijeka
  - University Hospital Center Split, Split
  - General Hospital Varazdin, Varaždin
  - Clinic for Tumors, Zagreb
  - University Hospital Center "Sestre milosrdnice", Zagreb
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Oncology Clinic, Medical center, Bezanijska Kosa, Belgrade

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991094&StudyName=Aromasin%AE%20As%20Adjuvant%20Treatment%20In%20Postmenopausal%20Women%20With%20Invasive%2C%20Estrogen%20Receptor%20Positive%20Early%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: Participants received exemestane (Aromasin) in accordance with Summary of Product Characteristics (SmPC) and adjusted according to medical and therapeutic necessity in a sequential adjuvant hormonal therapy (tamoxifen followed by Aromasin) up to 5 years or until tumor relapse occurred.
Period: Overall Study
Arm/Group | Exemestane
Started | 46
Completed | 0
Not Completed | 46
Not completed — Study terminated by sponsor | 45
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 59.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Type of Tumor [Number; unit: participants] — Number of participants with different types of tumor such as; ductal carcinoma, lobular carcinoma, invasive ductal carcinoma, invasive lobular carcinoma, papillary carcinoma, medullary carcinoma, mucinous (colloid) carcinoma and others.
  participants
    Invasive ductal carcinoma | 31
    Invasive lobular carcinoma | 7
    Papillary carcinoma | 0
    Medullary carcinoma | 1
    Mucinous (colloid) carcinoma | 2
    Other | 5
Type of Surgery [Number; unit: participants] — Number of participants who had undergone different type of surgeries which included mastectomy, axilla evacuation, breast quadrantectomy, dissectio axillae, radical mastectomy, axillary dissection, ablation of both breast, segmentectomy, lymphadenectomy, lumpectomy, core biopsy, sentinel lymph node biopsy, quadrantectomy, re-excision, tumorectomy.
  participants | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Hormone Receptor Status [Number; unit: participants] — Number of participants with positive estrogen receptors.
  participants | 46
Lymph Node Status [Number; unit: participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Tumor Node Metastasis (TNM) Stage [Number; unit: participants] — TNM:based on tumor size, if cancer cells had spread to nearby lymph nodes (LN), or distant (other parts of body) metastasis. Stages included:stage 0(no evidence of cancer cells), stage 1(T1N0M0), stage IIA(T0N1M0, T1N1M0, T2N0M0), stage IIB(T2N1M0, T3N0M0), stage IIIA(T0N2M0, T1N2M0, T2N3M0, T3N1orN2M0), stage IIIb( T4 anyNM0, any TN3M0),stage IIIC(any TN3M0), stage IV(anyT anyNM1), where T0=early form of tumor, T1=<2 centimeter(cm), T2=2-5 cm, T3=>2 cm, T4=large sized, N0=not spread to LN, N1=spread to 1 to 3,N2=spread to 4 to 9,N3=spread >10 axillary LN, M0=no metastasis, M1= Metastasis.
  participants
    Stage I | 18
    Stage IIA | 14
    Stage IIB | 5
    Stage IIIB | 4
    Stage IV | 0
    Stage IIIA | 4
    Stage IIIC | 0
    Other | 1
Histopathological Grade [Number; unit: participants] — The grade of a cancer depends on what the cells look like and the growth-rate. Lower grade indicates a slower-growing cancer and a higher grade indicates a faster-growing one. Grade 1 (resemble normal cells, not growing rapidly), grade 2 (grow faster than normal cells), grade 3 and 4 (abnormal cells, grow and spread aggressively).
  participants
    Grade 1 | 10
    Grade 2 | 19
    Grade 3 | 7
    Unknown | 10
Number of participants on chemotherapy [Number; unit: participants] — Number of participants who received chemotherapy. Chemotherapeutic drugs included doxorubicin, cyclophosphamide, docetaxel, fluorouracil, methotrexate , 5-fluorouracil, epirubicin, endoxan, farmorubicin, adriamycin, cytoxan, trastuzumab.
  participants | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Number of participants on radiotherapy [Number; unit: participants] — Number of participants who received radiotherapy as measured in radiations per centigray (Rads/cGy).
  participants | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Concomitant morbidities in the past [Number; unit: participants] — Participants who had a concomitant morbidity in the past; participants with more than one concomitant morbidity were counted for each of the concomitant morbidity classes applicable.
  participants
    Cholelithiasis | 1
    Intracranial aneurysm | 1
    Cystitis noninfective | 1
    Reproductive tract disorder | 3
    Hypertension | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness (to study drug) was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to Month 36
Population: Safety analysis set included participants who received at least one dose of the study medication during the observation period.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 46
participants | 2

2. Secondary Outcome: Number of Participants With Concomitant Morbidities
Description: Participants who had a concomitant morbidity during the study for any period of time; participants with more than one concomitant morbidity were counted for each of the concomitant morbidity classes applicable.
Time Frame: Baseline up to Month 36
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 46
participants
  Coronary artery disease | 1
  Glaucoma | 1
  Scotoma | 1
  Crohn's disease | 1
  Fatigue | 1
  Multiple allergies | 1
  Skin infection | 1
  Diabetes mellitus | 1
  Arthralgia | 2
  Collagen disorder | 1
  Intervertebral disc protrusion | 1
  Osteoporosis | 3
  Headache | 1
  Depression | 1
  Hypertension | 8

3. Secondary Outcome: Number of Participants With Concomitant Medications
Description: Concomitant medication (any medication other than, and in addition to, the study medication) taken for any period of time during the study and was coded by World Health Organization (WHO) medical dictionary.
Time Frame: Baseline up to Month 36
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 46
participants | 0

4. Secondary Outcome: Percentage of Participants Who Discontinued the Study Medication
Time Frame: Baseline up to Month 36
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Reasons for Discontinuation From Study Medication
Time Frame: Baseline up to Month 36
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Discontinuation
Time Frame: Baseline up to Month 36
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

7. Secondary Outcome: Recurrence-free Survival
Description: Recurrence-free survival defined as the time from the initiation of study medication to the date of confirmation of any recurrence - as local or distant breast cancer recurrence; new primary breast cancer (ipsilateral or contralateral), death due to any cause.
Time Frame: Baseline up to Month 36
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival
Description: Time in months from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 30.4. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death (up to Month 36)
Population: Data was not analyzed as the study was terminated due to insufficient number of participants enrolled in the study.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Exemestane
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 2/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=46)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Hot flush (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was prematurely discontinued, therefore not all data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.